CLINICAL TRIAL: NCT01749774
Title: Physical Activity and Testicular Cancer - a Pilot Study: Feasibility and Effects of a Program Including Information, Counseling and a Physical Activity Program for Patients With Testicular Cancer During and After Chemotherapy
Brief Title: Physical Activity and Testicular Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Gjensidigestiftelsen (Unknown); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Lene Thorsen, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011/2008a
Record Dates: First submitted 2012-11-30; First posted 2012-12-17 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Testicular Cancer
Keywords: Physical activity; Testicular cancer; Chemotherapy; Feasibility
MeSH Terms: conditions — Testicular Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity counseling (Experimental)
  Interventions: Behavioral: Physical activity counseling

INTERVENTIONS:
Behavioral: Physical activity counseling

SUMMARY:
The purpose of this study is to determine the feasibility and effect of a program including information, counseling and an individualized physical activity program on physical and psychological health during and after chemotherapy in patients with testicular cancer. It is hypothesized that the patients are able to complete the intervention with individual adjustments.

ELIGIBILITY:
Inclusion Criteria:

* Seminoma/non-seminoma
* Stage II-IV
* 3-4 BEP(bleomycin,etoposide and cisplatin)or 4 EP(etoposide and cisplatin)
* > 18 years
* Capable of reading and writing Norwegian

Exclusion Criteria:

* Conditions of a severity that contraindicate exercise without adjusted actions
* Mentally incompetent conditions
* Conditions of a severity that complicates the ability to participate in a supervised training program

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Muscle strength, 1RM (one-repetition-maximum) | Baseline (0 weeks), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in 1RM from baseline to post-intervention and follow-up

SECONDARY OUTCOMES:
Cardio respiratory fitness (VO2max) | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in VO2max from baseline to post-intervention and follow-up
Body composition (Lean body mass and fat mass) | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in body composition from baseline to post-intervention and follow-up
Metabolic disease markers (blood pressure, body mass index, glucose, high density lipoprotein cholesterol, triglycerides) | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in metabolic disease markers from baseline to post-intervention and follow-up
C-reactive protein (CRP) | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in CRP from baseline to post-intervention and follow-up
Creatinkinase (CK) | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in CK from baseline to post-intervention and follow-up
Creatinkinase - MB (CK-MB) | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in CK-MB from baseline to post-intervention and follow-up
Myoglobin | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in myoglobin from baseline to post-intervention and follow-up
Work status | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in work status from baseline to post-intervention and follow-up
Fatigue | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in fatigue from baseline to post-intervention and follow-up
Anxiety and depression | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in anxiety and depression from baseline to post-intervention and follow-up
Quality of life | Baseline (0 week), post-intervention (9-12 weeks) and follow-up (24 weeks)
  Change in quality of life from baseline to post-intervention and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lene Thorsen, PhD, Principal Investigator — Oslo universty hospital
Locations (1):
- Oslo university hospital, Oslo, Norway

REFERENCES:
- [Derived] Thorsen L, Kirkegaard C, Loge JH, Kiserud CE, Johansen ML, Gjerset GM, Edvardsen E, Hamre H, Ikdahl T, Fossa SD. Feasibility of a physical activity intervention during and shortly after chemotherapy for testicular cancer. BMC Res Notes. 2017 Jun 15;10(1):214. doi: 10.1186/s13104-017-2531-y. PMID 28619116